## UNIVERSITY OF HERTFORDSHIRE ETHICS COMMITTEE FOR STUDIES INVOLVING THE USE OF HUMAN PARTICIPANTS ('ETHICS COMMITTEE')

## FORM EC3 CONSENT FORM FOR STUDIES INVOLVING HUMAN PARTICIPANTS

| I, the undersigned [please give your name here, in BLOCK CAPITALS] |
|---|
| of [please give contact details here, sufficient to enable the investigator to get in touch with you, such as a postal or email address] |
| hereby freely agree to take part in the study entitled Biomarker Feedback on Health and Wellbeing and Exercise Adherence following a 6 Month Weight Management Course: A pilot Study |
| // III |

(UH Protocol number LMS/SF/UH/03620)

- 1 I confirm that I have been given a Participant Information Sheet (a copy of which is attached to this form) giving particulars of the study, including its aim(s), methods and design, the names and contact details of key people and, as appropriate, the risks and potential benefits, how the information collected will be stored and for how long, and any plans for follow-up studies that might involve further approaches to participants. I have also been informed of how my personal information on this form will be stored and for how long. I have been given details of my involvement in the study. I have been told that in the event of any significant change to the aim(s) or design of the study I will be informed, and asked to renew my consent to participate in it.
- **2** I have been assured that I may withdraw from the study at any time without disadvantage or having to give a reason.
- **3** In giving my consent to participate in this study, I understand that voice, video or photo-recording will take place and I have been informed of how/whether this recording will be transmitted/displayed.
- **4** I have been given information about the risks of my suffering harm or adverse effects. I have been told about the aftercare and support that will be offered to me in the event of this happening, and I have been assured that all such aftercare or support would be provided at no cost to myself. In signing this consent form I accept that medical attention might be sought for me, should circumstances require this.
- **5** I have been told how information relating to me (data obtained in the course of the study, and data provided by me about myself) will be handled: how it will be kept secure, who will have access to it, and how it will or may be used.
- **6** I understand that my participation in this study may reveal findings that could indicate that I might require medical advice. In that event, I will be informed and advised to consult my GP. If, during the study, evidence comes to light that I may have a pre-existing medical condition that may put others at risk, I understand that the University will refer me to the appropriate authorities and that I will not be allowed to take any further part in the study.
- 7 I understand that if there is any revelation of unlawful activity or any indication of non-medical circumstances that would or has put others at risk, the University may refer the matter to the appropriate authorities.
- **8** I have been told that I may at some time in the future be contacted again in connection with this or another study.

| Signature of participant | Date |
|-----------------------------------------|----------------------|
| Signature of (principal) investigator | Date |
| Name of (principal) investigator [in BL | OCK CAPITALS please] |
| DR LINDSAY BOTTOMS | |